CLINICAL TRIAL: NCT03606538
Title: A Phase I, Open Label, Study of 3,4-Methylenedioxymethamphetamine (MDMA) Tolerability and Pharmacokinetics in Subjects With Moderate Hepatic Impairment Compared to Matched Control Subjects With Normal Hepatic Function
Brief Title: MDMA in Subjects With Moderate Hepatic Impairment and Subjects With Normal Hepatic Function
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MPKH
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pharmacokinetics; Hepatic Impairment
Keywords: MDMA; metabolism; methylenedioxymethamphetamine; midomafetamine
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Matched group comparison of pharmacokinetics and metabolism of single dose of 80 mg MDMA in participants with moderate hepatic impairment and participants with normal hepatic function and matched on age, weight and gender.
Masking Description: No masking; open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate hepatic impairment (Experimental): Eight participants with moderate hepatic impairment receive a single dose of 80 mg midomafetamine HCl.
  Interventions: Drug: Midomafetamine HCl
- Normal hepatic function (Experimental): Eight participants, each matched on age, weight and gender to a participant with moderate hepatic impairment, receive a single dose of 80 mg midomafetamine HCl.
  Interventions: Drug: Midomafetamine HCl

INTERVENTIONS:
Drug: Midomafetamine HCl — 80 mg midomafetamine HCl
  Other Names: MDMA; 3,4-methylenedioxymethamphetamine; midomafetamine; MDMA HCl

SUMMARY:
The goal of this clinical trial to learn how MDMA is processed in people with abnormal liver function.

The main questions it aims to answer are:

Do people with abnormal liver function experience greater absorption of MDMA? Does the dose of MDMA need to be adjusted in people with abnormal liver function?

Researchers will compare people with abnormal liver function to people with normal liver function.

Participants will receive a single dose of MDMA then undergo periodic vitals measurements. They will remain at the study site for two more days undergoing more vitals measurements and having subjective effects and adverse events measured.

DETAILED DESCRIPTION:
This protocol is for a Phase 1, open-label study with a primary purpose of evaluating the effect of moderate hepatic impairment in the pharmacokinetics of MDMA and its active metabolite, 3,4-methylene-dioxyamphetamine (MDA), and determining whether an adjustment to the dosage would be indicated in this group of patients in comparison to patients with normal liver function. Because people with moderate hepatic impairment may experience greater exposure to drug than people without it, the secondary purpose of this study is to evaluate the effect of moderate hepatic impairment on the safety and tolerability of oral MDMA, with special attention to ECG data. The study will enroll eight participants, ages 18 to 65 years old, with moderate hepatic impairment, and eight healthy controls with normal hepatic function who are matched with participants with moderate impaired hepatic function on the basis of age, weight and gender.

Participants who give their written informed consent will be screened for study participation that will include a physical examination, assessing current and prior medical and physical health, and a baseline electrocardiogram (ECG) reading. If applicable, they may begin tapering off any contraindicated psychiatric medication. Participants who meet study criteria will receive a single dose of 80 mg midomafetamine HCl on the first day of a three-day stay at the study site.

Blood will be collected periodically in order to calculate pharmacokinetics of MDMA and its active metabolite methylenedioxyamphetamine (MDA). Blood will be collected ten times on Day 1 (-5 min, 0 hours (drug administration), 0.5 h, 1, 2, 4, 6, 7, 10 and 12 hours), starting five minutes before drug administration. Subjective effects of MDMA will be assessed through 15 visual analog scales at similar time points to blood collection, at 0.5, 1, 2, 4, 6 and 7 hours post-drug. There will be six 12-lead ECG measurements on Day 1.

Participants will remain at the study site for two more days. Drug safety will be assessed by measuring blood pressure, heart rate and body temperature after MDMA administrations, collecting adverse events throughout the study and measuring suicidal thoughts or behaviors with the Columbia Suicide Severity Rating Scale (C-SSRS). Blood will be collected 24 and 36 hours after drug administration, and ECG will be performed on Day 2, and a single ECG and blood draw will occur on Day 3, 4 and 5. Participants will return for eight and 15 days after drug administration. They will have a single blood draw on each day. The study ends 15 days after drug administration, approximately one month after screening.

The primary outcome measure will be area under the curve from dosing to last dose (AUC) of MDMA and MDA. AUC will be computed from plasma collected multiple times after a single dose of MDMA, twice on the day following the day of drug administration, and once daily for three more days. Other pharmacokinetic measures will be maximal values of MDMA and MDA (Cmax), and time to reach maximum MDMA and MDA levels (Tmax). Safety measures will also include a comparison of subjective effects across groups, ECG readings, number of adverse events, and suicidal ideation or behavior as measured via C-SSRS during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate hepatic impairment (class B according to Child- Pugh's criteria).
* Participants with normal hepatic function: no clinically significant findings from medical history, physical examination, laboratory values within protocol defined parameters.
* Age 18 to 65 years.
* Weight > 45 kg
* Negative Carbohydrate Deficient Transferrin blood test at Screening and negative breathalyzer alcohol test prior to trial drug administration.
* Negative urine test for drugs of abuse at Screening and prior to trial drug administration.
* Able to comprehend and willing to sign an informed consent form.

Exclusion Criteria:

* Have a current psychiatric diagnosis.
* Are pregnant or nursing, or are women of child bearing potential who are not practicing an effective means of birth control.
* Have acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within 2 weeks.
* Have autoimmune liver disease; esophageal variceal bleeding within 6 months prior to screening, unless successfully treated with banding, or gastric varices.
* Have spontaneous bacterial peritonitis within 3 months prior to screening.
* Have a portosystemic shunt, organ transplant, Wilson's disease, cholestatic liver disease (e g, primary biliary cirrhosis or primary sclerosing cholangitis)
* Evidence or history of significant hematological, endocrine, cerebrovascular, cardiovascular (including controlled hyper-tension), coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of MDMA administration.
* For moderate hepatic impairment participants: have clinically significant laboratory findings except as related to hepatic impairment.
* For control participants only: have clinically significant laboratory results outside the normal limits, including AST >48 U/L, ALT > 55 U/L, GGT > 48 U/L, bilirubin > 1.2 mg/dL or hemoglobin < 12 g/dL.
* Have a history of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject.
* Have any positive test for drugs of abuse and /or alcohol at screening.
* Have a history or presence of clinically significant abnormal 12-lead ECG or an ECG with QTc by Bazett's correction of > 450 ms in men, > 470 ms in women on the screening ECG.
* Have a PR interval > 240 ms, QRS > 110 ms or a history of prolongation of QT interval.
* Have mental incapacity, unwillingness or language barriers precluding adequate understanding or subject co-operation.
* Are unwilling to stay in the clinical unit for the required duration as per the protocol.
* Have a known or suspected allergy to trial product or related products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-03-29 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Area under curve from dosing time to last measurement (AUC(0-t)) - MDMA | 0 to 5 days after drug administration
  Computed exposure to MDMA using blood collected periodically at 1, 2, 4, 6, 7, 10, 12, 24, 36, 48, 72 and 96 h post drug
Area under curve from dosing time to last measurement (AUC(0-t) MDA | 0 to 5 days after drug administration
  Computed exposure to MDA using blood collected periodically at 1, 2, 4, 6, 7, 10, 12, 24, 36, 48, 72 and 96 h post-MDMA administration

SECONDARY OUTCOMES:
Peak MDMA (Cmax) | 0 to 5 days after drug administration
  Maximum value of plasma MDMA in nglml
Peak MDA (Cmax) | 0 to 5 days after drug administration
  Maximum value of plasma MDA in ng/lml
Time to maximum (Tmax) MDMA | 0 to 5 days after drug administration
  Time to reach maximum plasma values of MDMA
Time to maximum (Tmax) MDA | 0 to 5 days after drug administration
  Time to reach maximum plasma values of MDA
Area under curve from dosing time to infinity (AUC(0-infinity)) - MDMA | 0 to 5 days after drug administration
  Computed exposure to MDMA using blood collected periodically at 1, 2, 4, 6, 7, 10, 12, 24, 36, 48, 72 and 96 h post drug
Area under curve from dosing time to infinity (AUC(0-infinity)) - MDA | 0 to 5 days after drug administration
  Computed exposure to MDA using blood collected periodically at 1, 2, 4, 6, 7, 10, 12, 24, 36, 48, 72 and 96 h post drug
90% CL between hepatic impaired and no hepatic impairment groups for AUC (0-t) | 0 to 5 days after drug administration
  90% confidence interval (CI) for the ratio of population geometric means between moderate hepatic impairment and normal hepatic function for AUC (0-t)
90% CL between hepatic impaired and no hepatic impairment groups for AUC (0-infinity) | 0 to 5 days after drug administration
  90% confidence interval (CI) for the ratio of population geometric means between moderate hepatic impairment and normal hepatic function for AUC(0-infinity)
90% CL between hepatic impaired and no hepatic impairment groups for Cmax | 0 to 5 days after drug administration
  90% confidence interval (CI) for the ratio of population geometric means between moderate hepatic impairment and normal hepatic function for Cmax
Change in QTcI - Baseline to 0.5 h post drug | 0 days after drug administration
  Change in ECG QTcl from Baseline compared to 0.5 h post MDMA
Change in QTcI - Baseline to 2 h post-drug | 0 days after drug administration
  Change in ECG QTcl from Baseline compared to 2 h post MDMA
Change in QTcI Baseline to 4 h post-drug | 0 days after drug administration
  Change in ECG QTcl from Baseline compared to 4 h post MDMA
Change in QTcI Baseline to 6 h post-drug | 0 days after drug administration
  Change in ECG QTcl from Baseline compared to 6 h post MDMA
Change in QTcI Baseline to 7 h post-drug | 0 days after drug administration
  Change in ECG QTcl from Baseline compared to 7 h post MDMA
Change in QTcI Baseline to 1 d post-drug | 1 day after drug administration
  Change in ECG QTcl from Baseline compared to 1 d post MDMA
Change in QTcI Baseline to 2 d post-drug | 2 days after drug administration
  Change in ECG QTcl from Baseline compared to 2 d post MDMA
Change in QTcI Baseline to 3 d post-drug | 3 days after drug administration
  Change in ECG QTcl from Baseline compared to 3 d post MDMA
Change in QTcI Baseline to 4 d post-drug | 4 days after drug administration
  Change in ECG QTcl from Baseline compared to 4 d post MDMA
Pre-drug Systolic blood pressure (SBP) | 0 days after drug administration
  First SBP measurement, prior to drug administration, on day of drug administration
Peak Systolic blood pressure (SBP) | 0 days after drug administration
  Maximum value of SBP measured during day of drug administration
Final systolic blood pressure (SBP) | 0 days after drug administration
  Last SBP measurement taken on day of drug administration
Pre-drug Diastolic blood pressure (DBP) | 0 days after drug administration
  First DBP measurement, prior to drug administration, on day of drug administration
Peak Diastolic blood pressure (DBP) | 0 days after drug administration
  Maximum value of DBP measured during day of drug administration
Final Diastolic blood pressure (DBP) | 0 days after drug administration
  Last DBP measurement taken on day of drug administration
Pre-drug heart rate (HR) | 0 days after drug administration
  First HR measurement, prior to drug administration, on day of drug administration
Peak heart rate (HR) | 0 days after drug administration
  Maximum value of HR measured during day of drug administration
Final heart rate (HR) | 0 days after drug administration
  Last HR measurement taken on day of drug administration
Pre-drug body temperature (BT) | 0 days after drug administration
  First body temperature measurement, prior to drug administration, on day of drug administration
Peak body temperature (BT) | 0 days after drug administration
  Maximum BT value measured during day of drug administration
Final body temperature (BT) | 0 days after drug administration
  Last BT measurement taken on day of drug administration
Number of AEs reported | -4 days to 15 days post drug administration
  Number of AEs reported in each group from enrollment to study end

CONTACTS AND LOCATIONS:
Overall Officials: Janel Long-Boyle, PharmD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Alliance for Multispecialty Research, LLC., Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when all participants have completed the study
Access Criteria: Interested persons should correspond with the central contact for the multisite study.